CLINICAL TRIAL: NCT02573818
Title: Open-Label Post Approval Study of the SEDASYS System User Response to System Alarms
Brief Title: Sedasys Post Approval Study Users Response to System Alarms
Status: Terminated | Type: Observational
Why Stopped: franchise closed; no safety concerns
Sponsor: Ethicon Endo-Surgery (Industry)
Responsible Party: Sponsor
Other Study IDs: SED-14-001
Record Dates: First submitted 2015-10-06; First posted 2015-10-12 (Estimated); Last update posted 2017-03-24 (Actual); Status verified 2017-03

CONDITIONS: Conscious Sedation
Keywords: sedation for EGD and colonoscopy procedures

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- SEDASYS System
  Interventions: Device: SEDASYS System

INTERVENTIONS:
Device: SEDASYS System — propofol sedation with the SEDASYS System

SUMMARY:
The purpose of this study is to evaluate the users' responses to the SEDASYS® System alarms during esophagogastroduodenoscopy (EGD) or colonoscopy.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) I and II
* male and female
* Scheduled for routine colonoscopy or EGD
* ≥18 years of age
* Able to read, speak, and understand English

Exclusion Criteria:

* Physical or psychological condition which would impair trial participation, at the discretion of the PI
* BMI ≥ 35
* Pregnancy or lactation
* Known or suspected hypersensitivity to propofol or fentanyl
* Use of a fentanyl patch
* Allergies to eggs, egg products soybeans or soy products
* Diagnosis of sleep apnea
* Gastroparesis
* Full stomach at the time of procedure
* Participation in any other investigational device or drug study within 30 days of enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Male and female subjects 18 years or older scheduled for colonoscopy or EGD
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2015-09-01 (Actual); Primary Completion 2016-06-15 (Actual); Study Completion 2016-06-15 (Actual)

PRIMARY OUTCOMES:
Percent of documented responses/actions taken in response to SEDASYS System alarms (oxygen desaturation, apnea, hypotension, and bradycardia alarms) | <24 hours, i.e., for duration of study procedure

SECONDARY OUTCOMES:
Fraction of users responses/actions to oxygen desaturation, apnea, hypotension, and/or bradycardia alarms deemed sufficient by Endpoint Adjudication Committee (EAC) | assessment of sufficient alarms will be reviewed by EAC after 100, 400, and 866 subjects completed the study

CONTACTS AND LOCATIONS:
Overall Officials: James F Martin, PhD, Study Director — Ethicon Endo-Surgery, Inc.
Locations (1):
- ProMedica Toledo Hospital, Toledo, Ohio, United States

IPD SHARING:
Plan to Share IPD: No